CLINICAL TRIAL: NCT03069794
Title: Effect of Spinal Surgery on Stable Force Platform Parameters Estimating the Posture and the Balance of the Patients Reached of Spinal Pathologies
Brief Title: Effect of Spinal Surgery on the Posture and the Balance of the Patients Reached of Spinal Pathologies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STABILOMETRIE
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Spinal Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of stable force platform (Other): Ennrollment of every patient programmed for spinal surgery in orthopaedic service
  Interventions: Diagnostic Test: Use of stable force platform

INTERVENTIONS:
Diagnostic Test: Use of stable force platform — Use of stable force platform to appreciate the posture before and after spinal surgery

SUMMARY:
Many studies are in favour of the importance of the rachis on the postural balance of the body.It is possible to study the upright posture by determining the center of pressure using a platform of strength.The spinal surgery have two objectives ,mechanic and neurologic .By deformation correction and stabilizing vertebral stages via arthrodesis, it seems to hypothesize that surgery can modify postural balance.

This study aim to evaluate spinal surgery effect on posture using that plaftorm .

DETAILED DESCRIPTION:
At the inclusion, Day 1 and day 2 after surgery, the patient will stand on the stabilometric platform, with arms extended along the body, barefoot at 30 ° with a 2 cm gap at the heels.

He will fix a target located 1 meter away from him, in silence and will be instructed to "stand as still as possible, with his arms along his body, look in the direction of the visual target, do not think about anything. ". Then there will be a collection of data in 3 shots of 90 seconds, with a rest period between each shot, using the Winposture® software. The patient will answer health related quality of life questionnaires.

6 months after inclusion, patients will answer health related quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years old
* Patient programmed for spinal surgery
* Patient accepting participation

Exclusion Criteria:

* Refusal of participation
* All patient with vestibular disease
* All patient with neurologic disease
* Patient with pathologies not allowing to maintain the prolonged standing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2017-07-18 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
Center of foot pressure (COP) positions | Day 1- Day 2
  COP measurements by using stable force platform

CONTACTS AND LOCATIONS:
Overall Officials: Romain Clquin, Study Director — Groupe Hospitalier Paris St Joseph; Stéphane WOLFF, MD, Principal Investigator — Groupe Hospitalier Paris St Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided